CLINICAL TRIAL: NCT01210157
Title: GALectin-3 Binding Protein for Risk Assessment in Coronary arTery dIsease and Chronic Heart Failure
Brief Title: Galectin-3 Binding Protein in Cardiovascular Disease and Chronic Heart Failure
Acronym: GALACTIC
Status: Completed | Type: Observational
Sponsor: Heidelberg University (Other)
Responsible Party: Dr. Christian A. Gleissner, University of Heidelberg
Other Study IDs: GL_LGALS3BP
Record Dates: First submitted 2010-08-11; First posted 2010-09-28 (Estimated); Last update posted 2010-09-28 (Estimated); Status verified 2010-09

CONDITIONS: Heart Failure; Cardiomyopathies; Coronary Artery Disease
MeSH Terms: conditions — Heart Failure; Cardiomyopathies; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum, plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- I Ischemic CMP: Patients with impaired ventricular function caused by coronary artery disease.
- II CMP: Patients with impaired ventricular function which is not caused by coronary artery disease. Subgroups based on etiology (familial cardiomyopathy, toxic cardiomyopathy, etc.)

SUMMARY:
The purpose of this study is to determine whether galectin-3 binding protein plasma levels can predict adverse cardiovascular events in patients with coronary artery disease and/or heart failure.

DETAILED DESCRIPTION:
Chronic heart failure represents an important cause of disease burden in Western countries. Heart failure can be either caused by vascular disease (i.e. cardiomypathy (CMP) due to coronary artery disease ("ischemic/ICMP")) or by myocardial conditions (i.e. dilated cardiomyopathies (DCMP) resulting from other causes like familial disposition, drug toxicity, etc.). Gold standard for the diagnosis of CMPs is the coronary angiography in conjunction with left ventricular angiography and myocardial biopsy, non-invasive markers include C-reactive protein (CRP) for ICMP and brain natriuretic protein (BNP) for DCMP. We have previously identified G3BP to be overexpressed in foam cells and plasma-derived microparticles, both potentially important in formation of atherosclerotic plaque. Galectin-3 binding protein (G3BP) is a secreted protein that is involved in cell adhesion and immune activation. The purpose of the current study is to test, whether G3BP plasma levels (a) are able to non-invasively differentiate causes of CMP and (b) are a suitable means for future risk assessment in CMP patients.

ELIGIBILITY:
Inclusion Criteria:

* impaired ventricular function

Exclusion Criteria:

* neoplastic disease
* infections with hepatitis C or HIV

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing coronary angiography.
Sampling Method: Non-Probability Sample
Enrollment: 373 (Actual)
Dates: Start 2008-06; Primary Completion 2008-09 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Death from cardiac causes | up to five years

SECONDARY OUTCOMES:
diagnosis of coronary artery disease (CAD) | up to five years
diagnosis of cardiomypathy (CMP) | up to five years
assessment of disease stage (CAD-1-3, NYHA I-IV) | up to five years
non-fatal myocardial infarction or cerebrovascular accident | up to five years
revascularization (percutaneous coronary intervention (PCI) or coronary artery bypass graft (CABG)) | up to five years
rehospitalization | up to five years
implantation of ICD/biventricular pacemaker | up to five years
heart transplantation | up to five years
correlation with patient history | up to five years
correlation with physical examination | up to five years
correlation with routine lab values | up to five years
correlation with ECG | up to five years
correlation with echocardiography | up to five years
correlation with cardiac MRI | up to five years
correlation with cardiac CT | up to five years
correlation with chest X-ray | up to five years

CONTACTS AND LOCATIONS:
Overall Officials: Christian A Gleissner, MD, Principal Investigator — Heidelberg University
Locations (1):
- University of Heidelberg, Dept. of Cardiology, Heidelberg, Germany